CLINICAL TRIAL: NCT06939478
Title: vMap Informed Targeting of Arrythmia Location EP
Brief Title: AI Powered Mapping Technology for Identifying Arrhythmias
Acronym: VITAL-EP
Status: Recruiting | Type: Observational
Sponsor: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Collaborators: Vektor Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: VITAL-EP
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Data will be collected from participants who have previously been treated with the approved device as part of routine care.
  Interventions: Device: Arrhythmia Mapping
- Prospective: Data will be collected from participants prior to being treated with the approved device as part of routine care.
  Interventions: Device: Arrhythmia Mapping

INTERVENTIONS:
Device: Arrhythmia Mapping — vMap is indicated for analysis, display and storage of cardiac electrophysiological data and maps for analysis by a physician.

SUMMARY:
Exploratory, hypothesis-generating study evaluating the impact of vMap on procedural efficiency, acute success, and work flow optimization.

DETAILED DESCRIPTION:
The registry is a retrospective and prospective, post-approval, multicenter, single-arm, all-comers registry with two cohorts:

Retrospective Cohort: approximately 60 patients across two sites. Prospective Cohort: approximately 50 patients across two sites. This registry aims to collect real-world data on the clinical utility, safety, and procedural efficiency of vMap-guided ablation procedures.

ELIGIBILITY:
Retrospective Arm:

Inclusion Criteria:

1. Patients who had a standard of care cardiac ablation (de novo or repeat) where the vMap equipment was used.
2. The patient can provide written informed consent, if applicable.
3. The patient is greater than or equal to 18 years old

Prospective Arm:

Inclusion Criteria:

1. Patients who had a standard of care cardiac ablation (de novo or repeat) where the vMap equipment was used.
2. The patient can provide written informed consent, if applicable.
3. The patient is greater than or equal to 18 years old

Exclusion Criteria:

Participants who meet any one of the following criteria will be a screen failure and excluded from participation:

1. Non-inducible arrhythmia (unless pre-mapped via vMap prior to the procedure).
2. Patients in whom no ablation was performed using the vMap equipment.
3. Inability to obtain 12-lead ECG of sufficient quality for vMap analysis.
4. In the opinion of the Investigator, the participant is not suitable and has a contraindication to undergo the ablation procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be derived from subjects scheduled for cardiac ablation who meet inclusion and exclusion criteria for the registry.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AF Ablation rate of procedural efficacy | Day of procedure
  AF termination or AF non-inducibility in AF ablation cases
Focal Arrhythmia Ablation rate of procedural efficiency | Day of procedure
  Total procedure time, fluoroscopy time

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Grandview Medical Center, Birmingham, Alabama
  - Ascension St. Vincent's, Jacksonville, Florida
  - HCA Florida Healthcare, Miami, Florida
  - OhioHealth, Columbus, Ohio
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania